CLINICAL TRIAL: NCT04223661
Title: Frailty Score-guided Dosing of Lenalidomide, Dexamethasone and Daratumumab Induction Therapy in Elderly, Frail Newly Diagnosed Myeloma (MMY2035)
Brief Title: Frailty Score-guided Dosing of Lenalidomide, Dexamethasone and Daratumumab Induction Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Attaya Suvannasankha (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Indiana Institute for Medical Research (Other)
Responsible Party: Sponsor-Investigator, Attaya Suvannasankha, Assistant Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCC-0719
Record Dates: First submitted 2019-12-03; First posted 2020-01-10 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Intervention Model Description: Starting dose of lenalidomide in subjects who are intermediately fit (frailty score of 1) will be 10 mg day 1-21 of 28 day cycle and escalate to 15 mg, and in frail subjects (frailty score of 2 or higher) will be 5 mg, and escalate to 10 mg.
  All subjects will receive 20mg Dexamathasone and 1800mg Daratumumab during the course of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frailty score 1 (Experimental): Starting dose of lenalidomide in subjects who are intermediately fit (frailty score of 1) will be 10 mg day 1-21 of 28 day cycle and escalate to 15 mg
  All subjects will receive 20mg Dexamathasone weekly (split dosing is allowed) and 16mg Daratumumab (cycle 1-2 on days 1,8,15 and 22. Cycles 3-6 on days 1 and 15. Cycle 7 and beyond on day 1) during the course of the trial.
  Interventions: Drug: Lenalidomide Pill; Drug: Dexamethasone; Drug: Daratumumab
- Frailty Score 2 or above (Experimental): Starting dose of lenalidomide in frail subjects (frailty score of 2 or higher) will be 5 mg day 1-21 of 28 day cycle, and escalate to 10 mg.
  All subjects will receive 20mg Dexamathasone weekly (split dosing is allowed) and 16mg Daratumumab (cycle 1-2 on days 1,8,15 and 22. Cycles 3-6 on days 1 and 15. Cycle 7 and beyond on day 1) during the course of the trial.
  Interventions: Drug: Lenalidomide Pill; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Lenalidomide Pill — Lenalidomide will be administered PO on Days 1 through 21 of each 28 day cycle at the dose according to the frailty score and creatinine clearance.
Drug: Dexamethasone — Dexamethasone will be administered at 20 mg per week. During weeks when the subject receives an infusion of daratumumab, dexamethasone will be administered on infusion days at a dose of 20 mg IV before the infusion.
Drug: Daratumumab — Daratumumab (1800 mg) will be administered by SC injection by manual push over approximately 3 - 5 minutes in the abdominal subcutaneous tissues in the left/right locations, alternating between individual doses. The volume of the SC solution will be 15 mL for the 1800 mg dose

SUMMARY:
The purpose of this study is to determine if using a subject's baseline frailty score to guide the dosing of lenalidomide in a combination with dexamethasone and daratumumab (DRd lite).

DETAILED DESCRIPTION:
This is a multi-institution, prospective, single arm Phase II trial of lenalidomide in a combination with dexamethasone and daratumumab (DRd lite) with no blinding or randomization. This study will enroll 44 patients over 36 months.

Primary Objectives:

1. Evaluate Response rate
2. Evaluate Side effects

Secondary Objectives:

1. Evaluate Time on therapy
2. Evaluate Progression free survival
3. Evaluate Time to the next line of therapy
4. Assess Quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Newly diagnosed, symptomatic MM who have frailty score of 1 or higher; patients age ≥ 75 or younger patients with comorbidities (<75):

   Frailty score takes into account age, as well as the geriatric assessments incorporating 3 tools: the Katz Activity of Daily Living (ADL), the Lawton Instrumental Activity of Daily Living (IADL), and the Charlson Comorbidity Index (CCI)-see detailed tables in Appendix A.

   Score calculation tool: www.myelomafrailtyscorecalculator.net
3. ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2 within 14 days prior to registration.
4. Measurable disease according to the International Myeloma Working Group criteria:

   * Serum M-protein ≥1 g/dL
   * Urine M-protein ≥200 mg/24 h, or
   * Serum FLC (free light-chain) assay: involved FLC level ≥10 mg/dL provided serum FLC ratio is abnormal
   * Clonal bone marrow plasma cells ≥ 10%
5. No prior systemic therapy for myeloma is allowed. Surgery such as vertebroplasty or intramedullary rod placements, and local palliative radiation are allowed as long as subjects have no residual AEs (adverse events) from prior therapies at the time of screening
6. Life expectancy of >3 months as determined by the treating physician.
7. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 14 days prior to registration.

   System Laboratory Value Hematological* Absolute Neutrophil Count (ANC) ≥ 1.0 K/mm3 Platelet ≥ 50 K/mm3 Hemoglobin (Hgb) ≥ 8 g/dL Renal Calculated creatinine clearance ≥ 30 mL/min using 24 hour urine creatinine clearance Hepatic Bilirubin ≤ 2 × upper limit of normal (ULN) Aspartate aminotransferase (AST) ≤ 2 × ULN Alanine aminotransferase (ALT) ≤ 2 × ULN Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 2 × ULN
8. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
9. Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use one highly effective method of contraception and one barrier method from the time of informed consent until 3 months after treatment discontinuation. The birth control method must include one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy with confirmation of procedure) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap).
10. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Prior or concurrent exposure to any of the following:

   1. To daratumumab or other anti-CD-38 therapies
   2. Maximum of 40 mg dexamethasone (or equivalent) daily for a maximum of 4 days consecutively up to 21 days of 1st dose
   3. Exposure to investigational drug (including investigational vaccines) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer, before enrollment [Cycle 1, Day 1 / Randomization]
   4. Focal radiation therapy within 14 days prior to enrollmentrandomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma. Radiotherapy within 14 days prior to enrollmentrandomization on measurable extramedullary plasmacytoma is not permitted even in the setting of palliation for symptomatic management.
2. Known allergies, hypersensitivity, or intolerance to any of the study drugs, hyaluronidase, mannitol, sorbitol or, corticosteroids, monoclonal antibodies, human proteins, or their excipients.
3. Active infection requiring systemic therapy
4. Poorly controlled reactive airway diseases including COPD (chronic obstructive pulmonary disease) or asthma. In subjects with underlying disease of COPD or asthma, spirometric analysis is recommended. Subjects with FEV1 (forced expiratory volume at one second) < 50% is excluded.
5. Other medical conditions interfering with the administration of and compliance to treatments such as Cardiac disease (such as myocardial infarction within past 6 months, uncontrolled cardiac arrhythmia, congestive cardiac failure), major surgeries within past 2 weeks, plasmapheresis within past 28 days
6. Plasma cell leukemia or amyloidosis
7. Pregnant or breastfeeding
8. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
9. Active central nervous system (CNS) involvement by MM
10. Contraindication to receive antiplatelet or anticoagulant prophylaxis
11. Subject is:

    1. seropositive for human immunodeficiency virus (HIV)
    2. seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    3. seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-06 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 3 months
  Based on the International Myeloma Working group criteria
Response Rate | 6 months
  Based on the International Myeloma Working group criteria
Response Rate | 12 months
  Based on the International Myeloma Working group criteria
Response Rate | Best response achieved (up to but no longer than 2 years)
  Based on the International Myeloma Working group criteria
Side Effects | up to 730 days
  Evaluated based on CTCAE version 5.0

SECONDARY OUTCOMES:
Time on therapy | up to 730 days
  From the start of treatment till the end of treatment (of all 3 drugs)
Progression free survival | up to 730 days
  From the start of the treatment until the date of disease progression or death due to any cause. Subjects not progressing or dying will be censored at last disease evaluation date.
Time to the next line of therapy | up to 730 days
  Duration between the start of the study therapy of all 3 drugs and the start of any new line of therapy.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | Monthly (months 1-6), then every 3 months until treatment end (up to but no longer than 2 years)
  EORTC QLQ-C30
Quality of Life- Myeloma | Monthly (months 1-6), then every 3 months until treatment end (up to but no longer than 2 years)
  EORTC QLQ-MY20

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, MD, Principal Investigator — Indiana University
Locations (1):
- VA Roudebush Medical Center, Indianapolis, Indiana, United States